CLINICAL TRIAL: NCT07359534
Title: Recovery Following a Prolonged Period of Intensified Exercise Training: Evaluating the Impact of Levagen+® on Alleviating Physical, Physiological and Psychological Stress.
Brief Title: Training Health Recovery and Improvement Via Levagen+® Evaluation
Acronym: THRIVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Westminster (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Principal Investigator, Mohammed Gulrez Zariwala, Professor of Translational Physiology, University of Westminster
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: ETH2425-1214
Record Dates: First submitted 2026-01-12; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Exercise Recovery
Keywords: nutraceutical; exercise recovery; sport; cycling; inflammation; muscle recovery; sleep quality; Palmitoylethanolamide
MeSH Terms: conditions — Inflammation; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: double-blind, randomised
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levagen+® Palmitoylethanolamide (PEA) (Active Comparator): Levagen+® Palmitoylethanolamide (PEA) - 350mg/day, containing not less than 300 mg PEA
  Interventions: Dietary Supplement: Levagen+® Palmitoylethanolamide (PEA)
- Placebo (Placebo Comparator): Placebo - Microcrystalline Cellulose
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Levagen+® Palmitoylethanolamide (PEA) — Participants were instructed to consume 1 opaque capsule (350 mg Levagen+®, not less than 300mg PEA) with water daily at the same time of the day for 45 days.
  Arms: Levagen+® Palmitoylethanolamide (PEA)
Dietary Supplement: Placebo — Participants were instructed to consume 1 opaque capsule (Microcrystalline Cellulose) with water daily at the same time of the day for 45 days.
  Arms: Placebo

SUMMARY:
INTRODUCTION:

Sports supplements and ergogenic aids are widely used for performance enhancement in recreational and professional sports. Athletes undergo intense training to improve their cardiorespiratory and muscular systems, aiming for positive adaptations. However, intensified training without appropriate dietary support can pose risks such as inadequate muscle recovery, weakened immune function, and reduced sleep quality, leading to increased susceptibility to illness and heightened physiological and psychological stress. The recent removal of cannabidiol (CBD) from the World Anti-Doping Agency (WADA) prohibited list has increased its popularity among athletes for its potential benefits on recovery and sleep. However, concerns about its safety and legality in sport persist, leading many governing bodies to caution against its use.

Palmitoylethanolamide (PEA), a Generally Recognised as Safe (GRAS) supplement, exhibits anti-inflammatory effects and supports joint health. It also shows potential for stress and anxiety management, with ongoing research demonstrating this. Levagen+®, a formulated PEA, offers a safe, legal alternative to CBD, showing promise for recovery and sleep improvements. Additionally, PEA demonstrates neuroprotective and immunomodulating properties, indicating the potential benefits for athlete health, performance, and recovery. However, further research is needed to confirm Levagen+®'s efficacy as an ergogenic aid, especially in endurance sports.

The aim of this trial is to explore the effects of Levagen+® supplementation on physical, physiological and psychological recovery during a prolonged period (one week) of intensified cycling training, when administered over a period of 45 days.

DETAILED DESCRIPTION:
An intervention study with two treatment groups in a randomised, double-blind, crossover design.

Study population: Healthy, trained endurance cyclists (male or female) will receive supplements (active PEA or equivalent placebos allocated randomly) daily for 45 days, followed by a minimum 4-week washout period before receiving the other intervention.

Participants will be required to complete a cycling performance test (Functional Threshold Power [FTP] test) at home the day before attending laboratory testing visits 1, 2 and 4 (Day 0, Day 35 and Day 45 of supplementation), respectively. On the baseline first visit (Day 0), second (Day 35), third (Day 43) and endpoint fourth visits (Day 45) to the research facility, participants will be requested to complete an endurance cycling test (a 40 km time trial). Blood samples and pertinent questionnaires (Visual Analogue Scale (VAS) assessing muscle soreness; questionnaires assessing perception of exertion and arousal; sleep quality, mood and oral supplementation questionnaires) will also be collected at the aforementioned time points.

Participants will be required to follow and record their regular training regime from Day 1 to Day 35 of the study. The collected data over the course of these 5 weeks will be used to establish the intensified training protocol, whereby the average training load of the participant will be increased by 50%. The intensified training protocol will be assigned to participants to be completed over a 7-day period between the second visit (Day 35) and the third visit (Day 43). Participants will visit the research facility on Day 43 and Day 45 to assess recovery on day 1 and day 3 post intensified training period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Males and females (18-50 years of age)
* Trained cyclists/triathletes indicated by:
* Minimum functional threshold power (FTP, an indication of the highest average power output a cyclist can maintain for 60 minutes) of 2.9W/kg for males and 2.5W/kg for females
* Minimum 2 years of 5 hours cycling training a week

Exclusion Criteria:

* <18, >50 years
* Following a restrictive diet plan
* Consumption of >14 units of alcohol/week
* Allergies to test foods/drinks
* Illnesses or on medication (with a possible effect on taste and/or appetite)
* Devices such as pacemakers
* Smokers
* Gastrointestinal disorders
* Eating disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male and female
Enrollment: 20 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Exercise performance following intensified training during cycling tests in PEA supplemented athletes | The parameters will be measured before the 40km cycling time trial and every 10km during the trial (overall completion time will also be recorded) on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43), endpoint forth visit (Day45)
  The duration of completing the 40 km cycling time trial (hh:mm:ss)
Exercise performance following intensified training during cycling tests in PEA supplemented athletes | The parameters will be measured before the 40km cycling time trial and every 10km during the trial (overall completion time will also be recorded) on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43), endpoint forth visit (Day45)
  Perceptions of exertion (RPE: Borg 6-20 scale, where 6 equals no exertion and 20 equals maximal exertion)
Changes in levels of fatigue, quality of sleep, muscle soreness and mood during the intensified training and recovery period using questionnaires. | Questionnaires collected daily between days 33 and 45 (inclusive)
  Hooper and MacKinnon Questionnaire: a subjective assessment of the impact of DOMS in the domains of fatigue, sleep quality, general muscle soreness, stress level, and mood on a scale of 1-7, with higher scores denoting the worst results.
Changes in exercise-associated inflammatory markers associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Interleukin-6 (pg/mL)
Changes in exercise-associated inflammatory markers associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Tumour necrosis factor-alpha (pg/mL)

SECONDARY OUTCOMES:
Changes in exercise-associated oxidative stress markers associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Tbars (µM)
Changes in exercise-associated oxidative stress markers associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  F2-Isoprostane (pg/ml)
Changes in stress hormone levels associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Cortisol (nmol/l)
Changes in stress hormone levels associated with intensified training in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Testosterone (nmol/L)
Changes in neurotrophic factor levels in PEA supplemented athletes | The parameters will be measured before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Brain-Derived Neurotrophic Factor (pg/ml)
Perceptions of muscle pain associated with intensified training in PEA supplemented athletes | The parameters will be measured immediately before and immediately after exercise on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Visual Analogue Scale; scores range from 0 to 100 (the higher the score the greater the level of perceived pain)
Changes in state and profile of perceived mood during intensified training and recovery phase using questionnaires. | Questionnaires collected daily between days 33 and 45 (inclusive)
  Profile of Mood States (POMS) Questionnaire: a psychological assessment comprising forty questions. The forty items yield scores on six factors: Tension, Depression (depressed mood), Anger, Vigour, Fatigue, and Confusion. The responses are evaluated on five-point response scales ranging from 0 to 4, where 0 represents the 'lack of' and 4 represents the 'most extreme' experience of a particular feeling.
Perceptions of exercise-associated pleasure during endurance cycling (40km time trial) in PEA supplemented athletes | Perceived pleasure will be assessed immediately before the 40km time trial and every 10km during the trial, on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43) and endpoint forth visit (Day 45)
  Felt Arousal Scale: a 6-point Likert scale measuring arousal from 1 ("low arousal" to 6 ("high arousal").
Incidence and frequency of Levagen+® associated-gastrointestinal symptoms | gastrointestinal symptoms analysed daily during the supplementation period between days 33 and 45 (inclusive)
  Subjective analysis using the Gastrointestinal Symptoms Rating Scale (GSRS, on a 1 to 7 Likert scale, where 1 = no discomfort, 7 = very severe discomfort).
Metabolic changes following intensified training during cycling tests in PEA supplemented athletes | The parameters will be measured before the 40km cycling time trial and every 10km during the trial (overall completion time will also be recorded) on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43), endpoint forth visit (Day 45)
  Blood glucose concentration (mmol/L)
Metabolic changes following intensified training during cycling tests in PEA supplemented athletes | The parameters will be measured before the 40km cycling time trial and every 10km during the trial (overall completion time will also be recorded) on baseline first visit (Day 0), second visit (Day 35), third visit (Day 43), endpoint forth visit (Day 45)
  Blood lactate concentration (mmol/L)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gulrez Zariwala, PhD, Principal Investigator — University of Westminster
Locations (1):
- University of Westminster London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nerys Williams, The Borg Rating of Perceived Exertion (RPE) scale, Occupational Medicine, Volume 67, Issue 5, July 2017, Pages 404-405, https://doi.org/10.1093/occmed/kqx063
- [Background] J Wadley A, S Svendsen I, Gleeson M. Heightened Exercise-Induced Oxidative Stress at Simulated Moderate Level Altitude vs. Sea Level in Trained Cyclists. Int J Sport Nutr Exerc Metab. 2017 Apr;27(2):97-104. doi: 10.1123/ijsnem.2015-0345. Epub 2016 Oct 6. PMID 27710149
- [Background] Mallard A, Briskey D, Richards A, Mills D, Rao A. The Effect of Orally Dosed Levagen+ (palmitoylethanolamide) on Exercise Recovery in Healthy Males-A Double-Blind, Randomized, Placebo-Controlled Study. Nutrients. 2020 Feb 25;12(3):596. doi: 10.3390/nu12030596. PMID 32106527
- [Background] LoVerme J, La Rana G, Russo R, Calignano A, Piomelli D. The search for the palmitoylethanolamide receptor. Life Sci. 2005 Aug 19;77(14):1685-98. doi: 10.1016/j.lfs.2005.05.012. PMID 15963531
- [Background] Konopka AR, Harber MP. Skeletal muscle hypertrophy after aerobic exercise training. Exerc Sport Sci Rev. 2014 Apr;42(2):53-61. doi: 10.1249/JES.0000000000000007. PMID 24508740
- [Background] Kim N, Parolin B, Renshaw D, Deb SK, Zariwala MG. Formulated Palmitoylethanolamide Supplementation Improves Parameters of Cognitive Function and BDNF Levels in Young, Healthy Adults: A Randomised Cross-Over Trial. Nutrients. 2024 Feb 8;16(4):489. doi: 10.3390/nu16040489. PMID 38398813
- [Background] Killer SC, Svendsen IS, Jeukendrup AE, Gleeson M. Evidence of disturbed sleep and mood state in well-trained athletes during short-term intensified training with and without a high carbohydrate nutritional intervention. J Sports Sci. 2017 Jul;35(14):1402-1410. doi: 10.1080/02640414.2015.1085589. Epub 2015 Sep 25. PMID 26406911
- [Background] Kasper AM, Sparks SA, Hooks M, Skeer M, Webb B, Nia H, Morton JP, Close GL. High Prevalence of Cannabidiol Use Within Male Professional Rugby Union and League Players: A Quest for Pain Relief and Enhanced Recovery. Int J Sport Nutr Exerc Metab. 2020 Sep 1;30(5):315-322. doi: 10.1123/ijsnem.2020-0151. Epub 2020 Jul 30. PMID 32732454
- [Background] Keppel Hesselink JM, de Boer T, Witkamp RF. Palmitoylethanolamide: A Natural Body-Own Anti-Inflammatory Agent, Effective and Safe against Influenza and Common Cold. Int J Inflam. 2013;2013:151028. doi: 10.1155/2013/151028. Epub 2013 Aug 27. PMID 24066256
- [Background] Hellsten Y, Nyberg M. Cardiovascular Adaptations to Exercise Training. Compr Physiol. 2015 Dec 15;6(1):1-32. doi: 10.1002/cphy.c140080. PMID 26756625
- [Background] Gabrielsson L, Mattsson S, Fowler CJ. Palmitoylethanolamide for the treatment of pain: pharmacokinetics, safety and efficacy. Br J Clin Pharmacol. 2016 Oct;82(4):932-42. doi: 10.1111/bcp.13020. Epub 2016 Jun 29. PMID 27220803
- [Background] Evangelista M, Cilli, De Vitis R, Militerno A, Fanfani F. Ultra-micronized Palmitoylethanolamide Effects on Sleep-wake Rhythm and Neuropathic Pain Phenotypes in Patients with Carpal Tunnel Syndrome: An Open-label, Randomized Controlled Study. CNS Neurol Disord Drug Targets. 2018;17(4):291-298. doi: 10.2174/1871527317666180420143830. PMID 29676237